CLINICAL TRIAL: NCT00277017
Title: A Phase I/II Trial of Combination Therapy With 5-Fluorouracil, Interferon-an Interleukin-2, and Thalidomide for Metastatic, Advanced or Recurrent Renal Cell Carcinoma.
Brief Title: Combination Therapy With 5-Fluorouracil, Interferon-an Interleukin-2, & Thalidomide for Metastatic, Advanced or Recurrent Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1500C
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2009-12

CONDITIONS: Kidney; Cancer
Keywords: Combination Therapy; 5-Fluorouracil; Interferon-a Interleukin-2; Thalidomide; Renal Cell Carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; Interleukin-2; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 5-Flourouracil, Interferon-a, IL-2 and Thalidomide — Patients will receive oral dosages of Thalidomide at 200mg/day to start, with dosage gradually increasing up to a max of 1200mg/day. This will be taken in combination with:5-fluorouracil, given by continuous IV infusion over 24 hours (Day 1) every week for 4 weeks.
  Interferon-α, given subcutaneously on Day 1, 3 and 5 of every week for 4 weeks. Interleukin-2, given by continuous IV infusion Days 2-5, every week for 4 weeks.
  Treatment will be followed by 2 weeks of rest then repeated.
  Other Names: Flourouracil

SUMMARY:
The purpose of this study is to evaluate a therapy combining the established FUNIL regimen with Thalidomide. We want to see how well the therapy works, if it can be easily done, and how well the body handles the treatment. We also wish to see if the addition of Thalidomide will increase the effectiveness of the already established treatment regimen.

DETAILED DESCRIPTION:
Eligible patients who agree to take part in the study will receive oral dosages of Thalidomide at 200mg/day to start, with dosage gradually increasing up to a maximum of 1200mg/day. This will be taken in combination with:

5-fluorouracil, given by continuous IV infusion over 24 hours (Day 1) every week for 4 weeks.

Interferon-α, given subcutaneously on Day 1, 3 and 5 of every week for 4 weeks.

Interleukin-2, given by continuous IV infusion Days 2-5, every week for 4 weeks.

Treatment will be followed by 2 weeks of rest then repeated.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically proven renal cell carcinoma which is metastatic, non-resectable and/or recurrent.
* Patients must have bidimensionally measurable disease as defined in Section 10.1a documented within 28 days prior to registration. X-rays, scans, or physical exam of all non-measurable disease must be completed within 42 days prior to registration.
* Prestudy chest x-ray must be done within 42 days prior to registration.
* Prior treatment with drugs included in this protocol is permitted if such prior treatment occurred more than 6 months previous or if patient is currently exhibiting minor, mixed or partial response to any of these drugs. Prior treatment with other drugs is allowed as long as therapy was discontinued at least one month previously.
* Prior radiation therapy (to less than 25% of the bone marrow only, see section 19.2), or surgery are allowed. At least 4 weeks must have elapsed since the completion of radiation therapy, and there must be measurable disease outside the radiation fields. At least 3 weeks must have elapsed since completion of surgery.
* Patients must have had an EKG performed within 28 days prior to registration.
* Patients must have a Southwest Oncology Group performance status of 0-2 as defined in Section 10.4.

Exclusion Criteria:

* Patients must not be receiving or planning to receive concomitant biologic therapy, radiation therapy, hormonal therapy, or other chemotherapy while on this protocol (including G/GM-CSF).
* Patients with currently untreated brain metastases or brain metastases on current therapy are not eligible. Patients with prior brain metastases S/P radiation and/or surgery, and with stable response, confirmed by MRI, off corticosteroids may be eligible. Brain MRI within 28 days of treatment and consultation with the Study Coordinator is required for such patients.
* Pregnant or nursing women may not participate. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients with other serious illnesses, serious active infections requiring treatment with antibiotics, those requiring ongoing therapy with other investigational drugs or those receiving or expected to require corticosteroids are not permitted.
* Patients with known AIDS or HIV-1 associated complex or known to be HIV antibody seropositive are not eligible.
* In calculating days of tests and measurements, the day a test or measurement is done is considered Day 0. Therefore, if a test is done on a Monday, the Monday four weeks later would be considered Day 28. This allows for efficient patient scheduling without exceeding the guidelines. If Day 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day.
* Patients must be informed of the investigational nature of this study and give written in-formed consent in accordance with institutional and federal guidelines.
* Patients must be registered with the UNM Cancer Center Protocol Office. All records and flow sheets must be sent to this office.
* Active substance abuse can lead to unexpected and dangerous drug interactions and toxicities and impair compliance; therefore, this condition is an exclusion to registration or continuation on this study. Patients with a history of substance abuse must have blood or urine testing prior to registration on protocol. Psychosocial screening by the clinic psychologist or social worker is also suggested but not required. Patients found to be actively engaged in substance abuse while on protocol may be discontinued from protocol treatment at the direction of their physician and/or the study coordinator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Evaluate a therapy combining the established FUNIL regimen with Thalidomide. | Treatment stopped if there is disease progression or toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, MD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Lovelace Sandia Health Systems Dept of Hematology, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico